CLINICAL TRIAL: NCT03508362
Title: Neurobiological Substrate of Social Context on Cognitive Control in Drug Users
Acronym: STNdrugaddict
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-64; 2017-A03395-48 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Drug Use
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug user (Experimental): Regular use of cocaine
  Interventions: Device: Functional Magnetic Resonance Imaging (fRMI)
- Healthy volunteers (Active Comparator): non-drug user
  Interventions: Device: Functional Magnetic Resonance Imaging (fRMI)

INTERVENTIONS:
Device: Functional Magnetic Resonance Imaging (fRMI) — Acquisition of a functional MRI on the sub thalamic nucleus

SUMMARY:
The aim of the present project is to reveal, using Functional Magnetic Resonance Imaging (fMRI) in drug users, a specific modulation of brain structures and circuits involved in cognitive control (and especially those of inhibitory control) and reward while subjects are performing under the influence of drug-associated cues and in various social contexts.

This hypothesis, based on the animal work, is that the subthalamic nucleus (STN) should play a critical role in these processes. Addictive behaviour can be seen as a loss of control resulting from reduced inhibitory control, leading to compulsive drug use. These disorders are known to be associated with a hypoactivation of specific frontal regions such as the anterior cingulate cortex or the prefrontal cortex.

For the present experiment, it is chosen to use a procedure well established for neurophysiological and behavioural assessment of inhibitory processes : the " stop-signal reaction time task ".

This task requires to inhibit a motor response (press a button) at the onset of a stop signal (a tone) that occurs while the response is already engaged. In this task associated with fMRI, it was previously shown that the STN is involved in the control of inhibition. These results confirm our data in the rat, and especially those showing that STN lesions block the ability to stop. The stop signal task will thus be appropriate to study the effect of the social context on inhibitory processes in a population of cocaine users.

In cocaine abusers, it was shown that inhibitory processes are affected. Here we aim at testing this population of subjects while they perform the stop task, but adding an implicit cognitive load induced by visual cues associated or not with cocaine intake. Since it want to assess the influence of a peer on both the performance and the associated cerebral activities, it will also control the presence of a peer observer in the procedure.

There will thus be three experimental factors, one inter-subject factor (the experimental group, cocaine users or controls) and two intra-subject factors (cocaine associated or neutral cue; presence of a peer observer). The "stop-signal" task should induce increased activity of the STN that should be modulated by the cocaine-associated cues and by the presence of a peer.

ELIGIBILITY:
Inclusion Criteria:

Drug Users Group

* age between 18 and 65 years
* regular use of cocaine and crack
* willing to participate
* able to give consent
* not meeting any non-inclusion criteria
* right-handed

Healthy volunteers group

* age between 18 and 65 years
* non-drug user
* willing to participate
* able to give consent
* not meeting any non-inclusion criteria
* right-handed

Exclusion Criteria:

* protected persons
* lactating women
* intolerance to noise
* not a beneficiary of a social security scheme.
* no signature on the consent form
* significant psychiatric or neurological disorder
* known visual impairment and abnormal vision despite correction
* Contraindication to MRI examination
* Claustrophobia.
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
Functional MRI highlighting a specific modulation of the structures involved in the cognitive control circuit | 24 months
  Compare in each group the regional brain activity through the measurement of cerebral oxygenation (blood oxygenation level dependent, BOLD). Increased activity in the subthalamic nucleus (STN) in relation to drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No